CLINICAL TRIAL: NCT01693276
Title: Gemcitabine/Abraxane Chemotherapy and Dose Escalated Radiotherapy for Locally Advanced, Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Olugbenga Olowokure (Other)
Responsible Party: Sponsor-Investigator, Olugbenga Olowokure, Assistant Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCC-GI-01
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemzar/Abraxane and Radiation Therapy (Experimental): Patients will receive 2 cycles of gemcitabine and abraxane prior to the start of chemoradiation. Chemoradiation will commence 2 week after the completion of second cycle of gemcitabine/abraxane. Patients will receive an additional 2 cycles of gemcitabine and abraxane to start 2-4 weeks after the completion of chemoradiation. After the last two cycles of chemotherapy, if well tolerated with continued tumor response additional cycles of chemotherapy may be given.
  Interventions: Drug: Gemcitabine; Drug: Abraxane; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Gemcitabine — gemcitabine 1000mg/m2 given on day 1,8, and 15 of a 28 day cycle for 2 cycles prior to chemoradiation and post RT.
  Gemcitabine 450 mg/m2, 30-minute infusion, given weekly during chemoradiation for a total of 6 weeks.
  Other Names: Gemzar
Drug: Abraxane — Abraxane® 100 mg/m2 given on day 1,8, and 15 of 28 day cycle for 2 cycles prior to RT and each cycle post RT
  Other Names: nab-Paclitaxel
Radiation: Radiation Therapy — IMRT Dose escalation: 60 Gy (2 Gy/fraction)
  Other Names: RT

SUMMARY:
This study will analyze the effects, good and/or bad, of the drug Abraxane in combination with gemcitabine and gemcitabine with concurrent radiation therapy for patients with locally advanced pancreatic cancer that cannot be removed by surgery. All of the medications used in this study are FDA-approved for use in patients with pancreatic cancer.

DETAILED DESCRIPTION:
The long term goal is to improve survival of patients with unresectable pancreatic cancer. Additional potential benefits include increased probability of local control and decreased distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven carcinoma of the pancreas that is locally advanced
* ECOG performance status 0- 2
* Adequate labs
* No prior abdominal radiation therapy
* No other concurrent clinically evident malignancy, except inactive nonmelanoma skin cancer, inactive cervical cancer, or other cancer for which the patient has been disease-free for 5 years
* All disease must be encompassed within a radiotherapy portal
* Not pregnant or nursing

Exclusion Criteria:

* Patient has metastatic disease on radiological staging
* systemic therapy.
* Patient has known active infection with HIV, hepatitis C or hepatitis B
* Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
* Patient is deemed to be have obvious resectable disease at presentation
* Received any investigational agent within a month prior to enrollment.
* Neuroendocrine tumors of the pancreas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Increase overall survival | 23 months
  Estimated increase in median survival from 11 to 16 months

SECONDARY OUTCOMES:
Rate of local control | baseline to average up to 24 weeks
  Determine rate of local control from the date of start of treatment to the date of the time of local progression

CONTACTS AND LOCATIONS:
Overall Officials: Olugbenga Olowokure, MD, Principal Investigator — University of Cincinnati; Michelle Mierzwa, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States